CLINICAL TRIAL: NCT03408119
Title: Dried Plums Prevent Inflammation And Improve Bone Health in Osteopenic Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Bahram Arjmandi, Dr. Bahram H. Arjmandi, PhD, RD, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-05648
Record Dates: First submitted 2018-01-09; First posted 2018-01-23 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Osteoporosis, Osteopenia
Keywords: prune; dried plum; osteoporosis; osteopenia; men
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Multiple Endocrine Neoplasia Type 1 | interventions — Vitamin D; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): 100g daily dried plum consumption, plus 800 IU vitamin D and 450 mg elemental calcium
  Interventions: Dietary Supplement: Dried Plum; Dietary Supplement: 800 IU vitamin D and 450mg elemental calcium
- Group B (Experimental): 50g daily dried plum consumption, plus 800 IU vitamin D and 450 mg elemental calcium
  Interventions: Dietary Supplement: Dried Plum; Dietary Supplement: 800 IU vitamin D and 450mg elemental calcium
- Group C (Placebo Comparator): 800 IU vitamin D and 450 mg elemental calcium
  Interventions: Dietary Supplement: 800 IU vitamin D and 450mg elemental calcium

INTERVENTIONS:
Dietary Supplement: Dried Plum — Dried plum fruit, 100g or 50g depending on treatment group randomized to
  Arms: Group A; Group B
Dietary Supplement: 800 IU vitamin D and 450mg elemental calcium — Supplemental vitamin D and calcium to protect against further bone loss

SUMMARY:
The goals of this study are 1) to investigate the extent to which dried plum improves bone health by measuring bone density (a measure of bone strength) of whole body, hip, and forearm, indicators of bone formation and bone breakdown, and 2) to determine the anti-inflammatory effects of dried plum by assessing biomarkers of inflammation. Additionally, relevant medical history and lifestyle variables will be recorded.

DETAILED DESCRIPTION:
Osteoporosis in men is an important yet an understudied debilitating disease. To date, most therapies are directed towards postmenopausal osteoporosis, and the efficacy of these therapies is not established for male osteoporosis. Therefore, due to concerns regarding the increasing prevalence of male osteoporosis and minimal treatment options available, it is imperative to further investigate the role of readily available preventative therapies such as functional foods on improving bone health in men.

In general, consumption of fruits and vegetables has health-protective effects, in part, through the prevention of inflammation and its related conditions, including bone loss. These protective effects have been primarily attributed to their bioactive components, including polyphenols. Dried plums (Prunus domestica L.) have been ranked as having one of the highest oxygen radical absorbance capacities among the commonly consumed fruits and vegetables, likely due to the fact that they are a rich source of polyphenolic compounds, including chlorogenic acid and neochlorogenic acid, which are potent antioxidants. For these reasons, dried plums have been investigated to determine if they would have beneficial effects on bone health, and their bone-protective effects have been well-established in animal models and to some degree in humans by our laboratory as well as others.

The long-term goal of this proposed research is to develop new approaches to prevent chronic inflammation and subsequently to prevent and/or reverse bone loss in osteopenic men, thereby reducing the risk of osteoporotic fractures. The rationale for conducting this study is to test the extent to which dried plum prevents inflammation and improves bone health in osteopenic men. Based on the promising findings of our previous research studies and those of others, we hypothesize that chronic consumption of dried plum will prevent inflammation thereby preventing and/or reversing further bone loss at the lumbar spine in osteopenic men. Healthy men between the ages of 55 and 80 years old with a baseline lumbar spine bone mineral density (BMD) t-score between 1 and 2 standard deviations (SD) below the mean, characterizing mild to moderate bone loss, will be recruited. The study participants must not have been on drug therapy for osteoporosis and must not have begun a new exercise regimen known to affect bone metabolism for at least six months prior to the start of the study. Evaluation will be based on quantitative assessments of serum and urinary markers of bone formation and bone resorption and bone density measurements. Nutrition indices that are known to influence skeletal mass such as dietary intakes of calcium, protein, fiber, and magnesium will also be assessed as well as relevant medical history and lifestyle variables.

The rationale for selecting osteopenic men rather than those with normal bone is to test our hypothesis that dried plum reverses bone loss similar to male rats. However, no further loss of BMD should also be considered a positive finding. Men with a t-score < -2 SD will be excluded because they are close to being osteoporotic. Changes in BMD and bone mineral content (BMC) of the lumbar spine are the primary outcome variables. Secondary outcome variables are the changes in BMD and BMC of whole body, hip, and forearm; and biomarkers of inflammation and bone turnover. The rationale for choosing the lumbar spine as our primary outcome variable site, is due to the high rates of bone loss that typically occur first in the lumbar spine and other areas of high trabecular bone content where there are many metabolically active surfaces. To test our hypothesis, two specific aims are proposed as follows:

Aim 1: To investigate the extent to which dried plum improves bone health by measuring:

Aim 2: To determine the anti-inflammatory effects of dried plum by assessing:

Study Overview Two hundred men whose lumbar spine BMD t-score is between 1 and 2 SD below the mean will be recruited from primary care and specialty clinics and by advertisement at large. After an initial telephone screening, all participants will be requested to report to the study site for their first visit. On the first visit (screening), the Study Coordinator will provide the potential subjects with verbal and written explanation of the project and will answer any questions regarding the study. Then the individual will be asked to sign an informed consent form, followed by a DXA scan to confirm osteopenia. Baseline assessments will be performed for medical history, medications use, dietary intake, and physical activity. If volunteers meet the study criteria, they will be scheduled for their second visit two weeks later (actual baseline data collection) and randomly assigned to their treatment group: 50 g dried plum, 100 g dried plum, or control for one year. In order to provide some protection against further bone loss, all study participants will receive 500 mg elemental calcium and 400 IU vitamin D3 daily. They will be given a three-day food record to take home and bring back on the second visit. Additionally, subjects will be asked to collect a 24-hour urine sample the day prior to their next visit and bring this with them to the clinical research facility and they will repeat this the day prior to each subsequent visit. During each visit (baseline, 3, 6, and 12 months) between the hours of 6-10 A.M., venous blood will be drawn from the antecubital vein. Subjects' anthropometrics including height, weight, and waist and hip circumferences will be measured. Participants will be asked to complete a Physical Activity Questionnaire. Participants will undergo a DXA scan for bone density measurements (lumbar spine, whole body, hip, and forearm BMD and BMC) at screening (considered baseline for BMD and BMC values), 6 months, and 12 months.

Data Analyses - Descriptive statistics will be calculated for all variables and will include means, standard deviations, medians, minima and maxima. Distributions of outcome variables will be examined graphically for symmetry and for outliers. If a lack of symmetry is noted, the variable will be transformed before analysis, most probably by a logarithmic transformation. Extreme outliers will be investigated for technical or clerical errors. If the size of the measurement cannot be attributed to such an error, it will be included in the analysis and the effect of deleting the observation will also be reported. Baseline characteristics for the study groups will be compared and if differences occur in variables that could influence bone mass, subsequent analyses will adjust for the effects of these variables. The data will be analyzed using PC SAS version 9.3 and SAS PROC MIXED. The overall effect of treatments will be inspected. The primary outcomes of interest will be the changes observed in lumbar spine BMD and BMC from baseline. The secondary outcome variables will be change in hip, forearm, and total body BMD and BMC, and biochemical markers of bone formation and bone resorption. Some covariates such as initial bone mass and baseline characteristics identified in the preliminary analysis will be included. Other factors that might affect the results, such as physical activity, dietary intakes and ethnicity, will also be examined.

For statistical purposes, the study may be considered a factorial design (3 treatments)*(2 times) for density measurements and (3 treatments)*(4 times) for serum and urine analyses. It is a repeated measures on the time factor (2 levels for DXA and 4 levels for blood and urine analyses). Analysis of variance techniques appropriate for this design will provide the primary statistical hypothesis testing procedures. To directly address primary research questions, planned comparisons will be made between the changes from baseline in the control group with changes in the dried plum groups. These comparisons will be made using actual differences as response variable, with current values, values adjusted by covariance for baseline, and with change as % of baseline as response variable. Clearly these tests are not independent, but results may offer different insights. It is anticipated that some subjects may leave the study and dropout rates between the three groups; hence, Kaplan Myer time to event analysis will be used to examine for possible differences in time to dropout patterns. The comparison of changes will first be made using only data for subjects who finish the study. A second examination will be made as intent to treat analysis using the MIXED procedure to adjust for missing data.

The relationship between bone mass and biochemical markers of bone turnover will be investigated through linear correlation coefficients. The lumbar spine will be the primary site of interest although bone mass, i.e. BMD and BMC, at other sites will also be evaluated. Hip, forearm, and total body BMD and BMC, as well as serum and urinary biochemical indices of bone formation and resorption will comprise the secondary independent variables to be considered. Preliminary models will examine the effect of each biochemical index individually, and then stepwise methods of variable selection will be employed through the use of multiple regression models to determine which combination of indices is strongly associated with BMD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men, between the ages of 55 and 80, whose lumbar spine BMD t-score is between 0.1 and 2.5 SD below the mean will be included. Participants who are not on testosterone and/or other pharmacological agents known to affect bone, or who have initiated an exercise program within the past 12 months known to influence bone (e.g. resistance training exercise), will be enrolled in this proposed study.

Exclusion Criteria:

* The subjects who will be recruited for the study should not be receiving endocrine (e.g. prednisone, other glucocorticoids) or neuroactive (e.g. dilantin, phenobarbital) drugs or any drugs known to influence bone and calcium metabolism. Men who have initiated regular exercise regimens known to influence bone within the past 12 months prior to the study, e.g. resistance exercise training will also be excluded. Men whose BMD t-score at any site that falls below 2.5 SD of the mean will be excluded from the study. Furthermore, subjects treated with calcitonin, bisphosphonates, denosumab, raloxifene, anabolic agents, e.g. PTH and growth hormone, or steroids within a year prior to the start of the study will be excluded. In addition, subjects with metabolic bone disease, renal disease, cancer, cardiovascular disease, diabetes mellitus, respiratory disease, gastrointestinal disease, liver disease, or other chronic diseases will be excluded. Potential subjects with a body mass index (BMI) < 18 and > 40 will be excluded to avoid extremes in leanness/adiposity and to readily allow body composition assessment. If subjects smoke ≥ 20 cigarettes per day, they will be excluded. Also men who regularly consume dried plum or prune juice will not be accepted into the study.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men aged 55-80 with osteopenia in lumbar (L1-L4) vertebrae
Enrollment: 62 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Bone mineral density (spine) | 1 year
  BMD of the lumbar (L1-L4) vertebrae

SECONDARY OUTCOMES:
Bone mineral content (spine) | 1 year
  BMC of the lumbar (L1-L4) vertebrae
Bone mineral Density (other) | 1 year
  BMD of the ulna, hip, and total body
Bone Mineral Content (other) | 1 year
  BMC of the ulna, hip, and total body

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No